CLINICAL TRIAL: NCT01988428
Title: A Prospective Randomized Controlled Trial to Investigate the Effects of Training Emergency Medical Services (EMS) Personnel in Recognizing and Initiating Treatment in the Prehospital Setting Together With Early Administration of Antibiotics for Patients Suspected of (Severe) Sepsis and Septic Shock
Brief Title: Prehospital Antibiotics Against Sepsis Trial
Acronym: PHANTASi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Stichting Nuts Ohra (Other); Nederlandse Internisten Vereniging ( Dutch Association of Internists) (Unknown)
Responsible Party: Principal Investigator, Prabath W.B. Nanayakkara, Doctor, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL42001.029.13
Record Dates: First submitted 2013-11-05; First posted 2013-11-20 (Estimated); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Sepsis; Severe Sepsis; Septic Shock
Keywords: sepsis; severe sepsis; septic shock
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Ceftriaxone

STUDY DESIGN:
Masking Description: Open label
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard care (No Intervention): * standard care
  * training of ambulance personnel in recognizing sepsis and initiating pre-hospital treatment
- Antibiotics (Experimental): * ceftriaxone 2000 mg (after taking bloodcultures)
  * training of ambulance personnel in recognizing sepsis and initiating pre-hospital treatment
  Interventions: Drug: Ceftriaxone 2000 mg

INTERVENTIONS:
Drug: Ceftriaxone 2000 mg — Ceftriaxone 2000 mg
  Other Names: rocephin (roche)
  Arms: Antibiotics

SUMMARY:
Sepsis is one of the most frequent reasons for referral to emergency departments (EDs) worldwide. The incidence of sepsis is likely to rise in the upcoming years. Sepsis has a tendency to become more serious when left untreated with a high mortality rate, exceeding even those of myocardial infarction and stroke. Therefore, much effort has been put in to start with appropriate therapy as early as possible. Early goal-directed therapy (EGDT) in the emergency department with fluid resuscitation, administration of vasopressors/vasodilators and intravenous antibiotics in patients with severe sepsis and septic shock has indeed decreased mortality substantially. Emergency medical services (EMS) personnel have already made a significant difference in improving care for patients with acute coronary syndrome, multiple trauma and stroke. Patients with severe sepsis or septic shock could also benefit greatly from timely pre-hospital care. Earlier recognition and initiation of treatment by EMS personnel may improve survival even more.

Interestingly, the first hour of ED presentation seems to be the most critical hour. Administration of antibiotics and fluid resuscitation in the pre-hospital setting will reduce the time to administration substantially. In adults, to the best of our knowledge, no studies on the effect of pre-hospital administration of antibiotics have been performed. In children with meningitis, some uncontrolled studies show contradictory results, most probably due to bias by severity. We propose a non-blinded randomised multicentre clinical trial study on the efficacy of early, pre-hospital intravenous administration of broad spectrum antibiotics (ceftriaxone), which are effective against a wide variety of infectious pathogens that cause most common community-acquired infections) in patients referred to the ED with suspected severe sepsis or septic shock.

Objective: To evaluate whether early, pre-hospital administration of antibiotics, together with training of ambulance personnel in recognizing and initiating treatment reduces 28-day mortality in patients referred to the ED with suspected severe sepsis or septic shock

Study design: Non-blinded randomized multicentre clinical trial nested within a stepped wedge design

Study population: All patients above the age of 18 years, with suspected severe sepsis or septic shock and transferred to the ED by ambulance, are eligible for study inclusion

Intervention: prehospital antibiotics (ceftriaxone 2000 mg intravenously)

Main study parameters/endpoints: 28-day mortality, hospital length of stay, admission to intensive or medium care unit (ICU/MC), time to administration of antibiotics. Follow up of one year. QoL after one month after discharge.

DETAILED DESCRIPTION:
Introduction Sepsis is one of the most common and life-threatening diseases in the world, causing more deaths than AIDS, breast cancer and prostate cancer put together (8-10). Despite the fact that the mortality of sepsis is ten times higher than myocardial infarction and to five times higher than stroke, relatively little attention is given to sepsis (23-25). In recent years successful clinical care management pathways have been developed for patients suffering from a myocardial infarction, stroke or a trauma. Even though there is strong evidence in scientific literature to support the need for a series of time-dependent actions, for sepsis this is still not the case.

On 13 September 2012, the first ' World Sepsis Day ' was held with as main objective : 'to increase awareness for sepsis as a potentially lethal condition, which should be considered as a medical emergency ' (26). Prompt recognition and treatment are extremely important for improving survival, while patients who survive sepsis can still continue to suffer from physical or psychological symptoms. The likelihood and severity of these complications depends on a number of factors including the severity of sepsis and the length of stay in hospital stay and in ICU.

Definition Sepsis is defined as a proven or strongly suspected infection that is associated with a 'systemic inflammatory response syndrome ' (SIRS) (29,30). SIRS exists if at least two of the four criteria are met: abnormal body temperature, increased heart rate (over 90 beats per minute), increased respiratory rate (more than 20 per minute) and an abnormal white blood cell (WBC) count. There are different degrees of sepsis on the basis of severity. Sepsis may develop to severe sepsis or septic shock, if treatment is not timely initiated. Severe sepsis is defined as sepsis with failure of one or more organ systems and septic shock and severe sepsis with persistent low blood pressures despite adequate resuscitation. In particular organ failure and shock cause high mortality.

In the Netherlands, more than 10,000 patients with sepsis are admitted to a hospital annually, with an average length of stay (LOS) of 15 days. The medical costs being approximately $ 20,000 per person, the total cost of severe sepsis in the Netherlands is estimated at nearly 170 million per year (1-3).

Mortality can be very high if sepsis is not timely or adequately treated, especially among the vulnerable elderly population. The mortality rates vary from 20 to 60 percent, depending on the age and other underlying diseases such as diabetes and cancer. Even in the VUmc the mortality rates are almost up to 40%. Multiorgan failure due to sepsis and septic shock is the leading cause of death in the ICU (31,32). The incidence of sepsis has increased in recent years and it is expected that this trend will continue, partly due to the aging population and partly because of increasing numbers of immune-compromised patients who are highly susceptible to all kinds of (opportunistic) infections.

Early Goal Directed Therapy (EGDT)

The advent of antibiotics was a major step forward in the treatment of sepsis, causing a mortality decrease by approximately 25 percent (33,34). It is noteworthy that in the decades hereafter very little progress in the treatment of sepsis was made, until the introduction of the 'Early goal directed therapy (EGDT). A study by Rivers and colleagues (4) shows that by applying EGDT during the first six hours after detection of sepsis, an absolute mortality reduction of almost 16% is achieved. This EGDT consists of a number of interventions, which have the purpose to optimize hemodynamics as quickly as possible by means of tight monitoring of arterial / venous pressures and oxygen saturation. The cornerstones of this treatment include aggressive fluid resuscitation, administration of vasopressors, giving protective ventilation and administration of broad-spectrum antibiotics. Several large clinical trials have confirmed the value of EGDT with sometimes even greater mortality reduction (35-38).

Survival Sepsis Campaign Timely recognition and rapid treatment of sepsis appears crucial, but recognizing sepsis still remains a challenge: the symptoms are often non-specific and various other diseases might fit as well. Therefore the "Surviving Sepsis Campaign" (SSC) was launched in 2003 (13), with the aim of creating awareness for sepsis for better recognition and treatment of sepsis to improve the prognosis. Through this campaign a directive was developed wherein a somewhat modified form of the EGDT was incorporated. This directive also states that broad-spectrum antibiotics should be administered as soon as possible, preferably within one hour after arrival in the emergency room.

Despite extensive attention in the last few years (major campaigns of VMS) in shortening time to administration of antibiotics (the so called "onset to needle time"), there are still delays in the start up of antibiotic therapy in the emergency department (ED) (6-7). EDs are still not functioning optimally, with waiting times sometimes exceeding 6 hours. This is also the conclusion of the report: 'Haastige spoed niet overal goed' from 2004 (Inspectie der Volksgezondheid). Herein EDs in the Netherlands are described as the weakest link in the emergency care, and in addition according to this report, little progress in the quality of care in the emergency department was made from 1994 to 2004. After much effort and recommendations, progress was made in the last few years but not sufficiently enough (see report '' Ziekenhuizen goed op weg met implementatie normen voor afdelingen spoedeisende hulp' "). Our study will therefore be able to contribute to the improvement of both in-hospital and pre-hospital acute care chain. Not only will we save costly time in the trip till reaching the hospital, but moreover we will also overcome (potential) delays in the emergency department by starting therapy in the ambulance. Delays which can amount from one to even six hours.

Why antibiotics should be administered early? The first hour of presentation in the emergency room, also known as the 'Golden Hour' seems to be the most critical one in the treatment of a septic patient. Retrospective studies have shown that rapid antibiotic administration could mean better chance of survival as well as a reduction in the chance of lasting physical problems. Moreover, rapid intervention may shorten hospital stay as well and even prevent the need for ICU admission (1-5). In daily practice however, implementation of the SSC directives is not always easy, and there may be several reasons to delay the start of treatment (6.15). The so-called 'onset to needle time' can be as high as several hours. A recent pilot study in the VUMC showed that 25% of patients had to wait longer than three hours at the emergency department before treatment was initiated with antibiotic therapy (16). Not only in the pilot study of our university but also in a retrospective study conducted by Kumar and colleagues only 32.5% of the patients received the first gift within the first 3 hours (6) Any delay in the administration of antibiotics, causes an increase in mortality rate with almost 8 percent per hour!(6).

The later the treatment is initiated, the greater the chance of multiorgan failure. Besides higher mortality-rates, multiorgan failure is directly correlated with more complications, longer hospital stay and higher use of costly healthcare facilities (10). Therefore it is probably important that the onset to needle time is as short as possible.

Moreover in the long term sepsis can cause much damage (17-20). Patients who survive sepsis often suffer for months of complications that arise during or after a prolonged hospitalization in intensive care (eg. critical illness neuropathy, problems with speech or swallowing by prolonged ventilation). The quality of life can also sharply deteriorate after experiencing sepsis (18).

An important point to note is that all the studies which state that early antibiotic administration is associated with improved survival, were retrospective and uncontrolled studies, making occurrence of selection bias probable. One of the reasons why the doctors may not be very keen on initiating the antibiotics early (before a definitive diagnosis is made) may be the fact that they consider current evidence insufficient and incomplete. In order to investigate the optimal timing of antibiotic administration, prospective randomized controlled studies should be performed at the emergency department. However, it may be unethical to randomize patients and delay initiation of antibiotic therapy at the ED. An alternative and perhaps a better option is to perform a prospective randomized trial in the pre-hospital setting, i.e in the ambulances. In current practice, initiation of antibiotic therapy starts at the emergency department (ED) and not in the ambulances. Pre-hospital antibiotic administration on the one hand may be a solution to avoid delays in treatment at the ED and on the other hand a way to finally perform a randomised trial to examine the effect of onset to needle time on clinical endpoints such as improved survival, shorter hospital stay and better quality of life.

Pre-hospital care, even in sepsis? Ambulance personnel have already made a significant contribution in improving care for patients with acute coronary syndrome, stroke and multiple trauma (42, 43). Patients with severe sepsis or septic shock can also benefit from early pre-hospital care (44). Pre-hospital care is the initial medical care, which is given by ambulance personnel once they reach the patient. Since time plays a crucial role in the treatment of sepsis, early recognition and initiation of treatment by the ambulance personnel may help to reduce mortality. The provision of pre-hospital care is associated with a shorter start-up time of EGDT and antibiotic therapy in the hospital (44-47). In addition, it appears that this pre-hospital care leads to quicker achievement of an optimal blood pressure, and oxygen saturation. Therefore, it can be expected that by the administration of broad-spectrum antibiotics in the ambulance, the survival of sepsis can be improved by greatly reducing the time to the administration of the necessary antibiotics.

To date no randomized controlled trials on the effect of antibiotics in the pre-hospital settings on adults have been conducted. In children with meningitis some uncontrolled studies have been done. In the studies by Strang and Cartwright (50,51), a clear beneficial effect on survival is seen after pre-hospital administration of antibiotics by general practitioners. Hamden and Sorensen (52.53) on the contrary showed that administration of antibiotics in the pre-hospital setting was associated with worse outcomes. A possible explanation for these divergent results is that there occurred a strong selection bias. The group of children receiving pre-hospital antibiotics could be in a more critical stage of illness.

A definitive answer to the question whether administration of antibiotics in pre-hospital setting is effective, can only be obtained by a prospective randomized controlled trial. In this form of study selection bias can be avoided.

However, recognition of sepsis is difficult, Suffoletto et al investigated how accurately the ambulance personnel in Pennsylvania were able to recognize a serious infection, the negative predictive value was 93%. In contrast, 69% of the patients with a severe infection were missed (8). A pilot study in Maastricht showed (54), that this situation can probably be extrapolated to the Netherlands as well: a large proportion of patients with septic shock was in fact not recognized as such and transported with a B-ride (low priority ride). The information transfer is hereby often incomplete or not entirely accurate (from the general practitioner to the ambulance personnel/hospital or from the ambulance to the ED) causing substantial delays in initiating treatment. Therefore, much can be gained by training ambulance personnel and getting them skilled enough in recognizing sepsis and improving the transfer of information.

Research Consortium

Through an intensive collaboration of some major Dutch medical centres and ambulance services, a research consortium has been established to start a nationwide project in the form of a multicentre randomized trial: the PHANTASi trial (PreHospital ANTibiotics Against Sepsi) This consortium has a joint goal namely evaluating the effect of early administration of antibiotics in patients with suspected sepsis in the pre-hospital setting compared to that with the regular treatment. Our hypothesis in this study is that administration of antibiotics in the pre-hospital setting will significantly shorten the time to administration of antibiotics, which subsequently will lead to improved survival. In addition, the pre-hospital administration of antibiotics shortens hospital stay which, simultaneously has a favorable effect on the cost and quality of life (QoL).

Importance of this project Sepsis is a major global health problem with an increasing incidence and high mortality rate. While in the past decades, modern medicine has become increasingly sophisticated, and the treatment and care around diseases, such as heart failure and cancer is greatly improved, treatment of sepsis remains a problem with a high mortality. Early administration of antibiotics in critically ill patients with sepsis could possibly change that. It is not clear what the best time of administration should be, because how early is early? Moreover, in practice it often happens that the time limits are not, or not sufficiently monitored closely, whilst increasing the risk of death.

Moreover, the treatment of an acutely ill patient requires teamwork and an optimally functioning acute-care chain. Through this project it will be possible to investigate whether pre-hospital antibiotic therapy leads to better outcomes for this category of seriously ill and vulnerable patients.

REFERENCES

1. van Gestel et al. Prevalence and incidence of severe sepsis in Dutch intensive care units. Critical Care August 2004, Vold 8 No 4
2. Roedig A (RIVM). Ziekenhuisopnamen sepsis en pyemie 2001-2004. In: Volksgezondheid Toekomst Verkenning, Nationaal Kompas Volksgezondheid. Bilthoven: RIVM
3. J. Bakker, et al Sepsis, een gecompliceerd syndroom met belangrijke medische en maatschappelijke consequentiesNedTijdschrGeneeskd. 2004;148:975-8
4. Rivers E, et al. Early goal-directed therapy in the treatment of severe sepsis and septic shock. NEJM. 2001; 345(19):1368-77.
5. Gaieski et al. Impact of time to antibiotics on survival in patients with severe sepsis or septic shock in whom early goal-directed therapy was initiated in the emergency department. Crit Care Med. 2010 Apr;38(4):1045-53.
6. Kumar et al. Duration of hypotension prior to initiation of effective antimicrobial therapy is the critical determinant of survival in human septic shock. Crit Care Med. 2006;34(6):1593
7. Vegting et al. Analysing completion times in an academic emergency department: coordination of care is the weakest link. The Netherlands Journal of Medicine. 2011 Sep; 69(9):392-398
8. Angus DC, et al. Epidemiology of severe sepsis in the United State: Analysis of incidence, outcome, and associated costs of care. Crit Care Med 2001;29(7)1303
9. Martin GS, et al. The epidemiology of sepsis in the United States from 1979 through 2000.NEJM. 2003;348:1546-54.
10. Vincent JL, Set al. Sepsis Occurrence in Acutely Ill Patients Investigators. Sepsis in European intensive care units: results of the SOAP study.Crit Care Med. 2006 Feb;34(2):344-53.
11. Kumar G et al . Nationwide trends of severe sepsis in the 21st century (2000-2007). Chest, 2011. 140(5): p. 1223
12. http://www.vmszorg.nl/10-Themas/Sepsis
13. Dellinger RP, et al. Surviving Sepsis Campaign: International guidelines for management of severe sepsis and septic shock: 2008. Crit Care Med 2008; 36:296 -327.
14. Tromp et al. The effects of implementation of the surviving sepsis Campaign in the Netherlands
15. O'Neill et al. Early goal directed therapy (EGDT( for severe sepsis/septic shock: which components of treatment are more difficult to implement in a community based emergency department?. The journal of Emergency Med.Vol 42, No5
16. Wetenschappelijk stage: S.B van der Meer, P.W.B. Nanayakkara, E.Schrijver Diagnostics of patients with sepsis or septic shock at the Emergency Department: Factors contributing to the delay of timely Administration of Antibiotics. Departments of Emergency Medicine and Internal Medicine, VU University Medical Centre Amsterdam, The Netherlands
17. Lazosky et al. Quality of life after septic illness. Journal of Critical Care (2010) 25 406-412
18. Hofhuis et al. The impact of severe sepsis on Health-Related quality of life: A long term follow-up study. Vol 107. No 6 Dec 2008
19. Iwashyna TJ, Ely EW, Smith DM, et al.: Long-term cognitive impairment and functional disability among survivors of severe sepsis. JAMA, 304: 1787-1794, 2010.
20. Oeyen et al. Quality of life after intensive care: A systematic review of the literature . Crit Care Med 2010 Vol 38. No 12
21. Siddiqui S, Razzak J. Early versus late pre-intensive care unit admission broad spectrum antibiotics for severe sepsis in adults. Cochrane Database of Systematic Reviews 2010, Issue 10.
22. http://acuteinterne.medconinternational.com
23. Yeh RW et al Population trends in the incidence and outcomes of acute myocardial infarction. N Engl J Med, 2010. 362(23): p. 2155-65.
24. Feigin et al, ; Worldwide stroke incidence and early case fatality reporten in 56 population based studies: a systematic review.
25. Ron Daniels, Surviving the first hours in sepsis: getting the basics right (an intensivist's perspective) J Antimicrob Chemother 2011; 66 Suppl 2: ii11-ii23
26. http://world-sepsis-day.org
27. Rattray JE, Johnston M, Wildsmith JA. Predictors of emotional outcomes of intensive care. Anaesthesia 2005;60:1085-92.
28. Hall MJ et al, Inpatient care for septicemia or sepsis: A challenge for patients ands hospitals. NCHS data brief, no 62, Hyattsville, MD: National center for Health statistics, 2011
29. Levy M et al. 2001 SCCM/ESICM/ACCP/ATS/SIS International Sepsis Definitions Conference. Crit Care Med 2003;31(4):1250-56
30. Bone RC. Definitions for sepsis and organ failure and guidelines for the use of innovative therapies in sepsis. Chest 1992;101:1644.
31. Balk RA. Pathogenesis and management of multiple organ dysfunction or failure in severe sepsis and septic shock. Crit Care Clin. 2000;16:337-52, vii.
32. Mayr VD et al. Causes of death and determinants of outcome in critically ill patients .Crit Care. 2006;10(6) :R154
33. Anand Kumar, Optimizing Antimicrobial Therapy in sepsis and septic shock. Crit Care Clin 25 (2009) 733-751.
34. Hemminki E, Paakkulainen A. Effect of antibiotics on mortality from infectious diseases in Sweden and Finland. Am J Public Health 1976;66:1180-4.
35. Sivayoham et al. Outcomes from implementing early goal-directed therapy for severe sepsis and septic shock: a 4 year observational cohort study. EJEM 2012, Vol 19 No 4
36. Rivers et al, Early interventions in severe sepsis and septic shock: a review of the evidence one decade later. Minerva Anestiol.2012; 78:712-2
37. Shapiro et al. A blueprint for a sepsis protocol. Acad Emerg Med April 2005, Vol.12, No 4
38. Jones AE et al. The effect of a quantitative resuscitation strategy on mortality in patients with sepsis: a meta-analysis. Crit Care Med 2008; 36: 2734-2739
39. hutchison
40. Barlow et al. Reducing door to antibiotic time in community-acquired pneumonia: controlled before and after evaluation and cost-effectiveness analysis. Thorax. 2007; (62 (1): 67-74
41. vanTuijn et al. Reduction of the onset to needle time for administration of antibiotics in patients with a severe infection: a tailored intervention project.Neth. Journal of Medicine, march 2010, Vol.68 no 3
42. Ghosh and Pepe, 2009 The critical care cascade: a systems approach. Current opinion in Critical Care, 15:279-283
43. Robson et al 2009 Sepsis: a need for prehospital intervention?.Emerg Med J, 26:535-538
44. Seymour et al, 2011. Understanding of sepsis among emergency medical services: a survey study. The Journal of Emergency Medicine, 1-12
45. Studnek et al, 2012. The impact of emergency medical services on the ED care of severe sepsis. The American Journal of Emergency Medicine, 30: 51-56
46. Band et al, 2011. Arriving by Emergency Medical Services improves time to treatment endpoints for patients with severe sepsis or septic shock. Academic Emergency Medicine, 18:934-940
47. Seymour et al,Out-of-hospital fluid in severe sepsis: effect on early resuscitation in the emergency department. 2010. Prehospital Emergency Care, 14:145-152
48. Proulx et al. Delays in the administration of antibiotics are associated with mortality from adult acute bacterial meningitis. Q J Med 2005; 98:291-298
49. Miner et al. Presentation, time to antibitotics and mortality of patients with bacterial meningitis at an urban county medical center. J of Emergency Med. Vol 21. No4, pp387-392, 2001
50. Cartwright K, Strang J, Gossain S, Begg N. Early treatment of meningococcal disease. BMJ 1992; 305(6856):774.
51. Strang JR, Pugh EJ. Meningococcal infections: reducing the case fatality rate by giving penicillin before admission to hospital. BMJ 1992;305:141-3. (18 July.)
52. Sorensen HT, Nielsen GL, Schonheyder HC, Steffensen FH, Hansen I, Sabroe S et al. Outcome of pre-hospital antibiotic treatment of meningococcal disease. J Clin Epidemiol 1998; 51(9):717-721.
53. Harnden A, Ninis N, Thompson M, Perera R, Levin M, Mant D et al. Parenteral penicillin for children with meningococcal disease before hospital admission: case-control study. BMJ 2006; 332(7553):1295-1298
54. Groenewoudt M, Roest AA, Leijten FM, Stassen PM ; .Eur J Emerg Med. 2013 Nov 6

ELIGIBILITY:
Inclusion Criteria:

- All patients older than 18 years who are suspected of sepsis AND have an abnormal temperature (>38 degrees Celsius or < 36 degrees Celsius) in combination with at least one of the following two SIRS criteria, abnormal pulse (> 90 beats per minute) and/or abnormal respiratory rate (> 20 per minutes)

Exclusion Criteria:

* Age <18 years
* Known severe allergic reaction to ceftriaxone or to other beta lactam antibiotics
* Known pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2672 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
mortality | 28 day mortality
  To evaluate whether early, pre-hospital administration of antibiotics reduces 28-day mortality in patients referred to the ED with suspected severe sepsis or septic shock.

SECONDARY OUTCOMES:
length of stay | an expected average of 5 weeks
  To compare whether there is a difference in the length of hospital stay in the standard treatment group versus the intervention group.

OTHER OUTCOMES:
quality of life | one month after discharge hospital
  To evaluate whether early antibiotic administration has a beneficial effect on the quality of life after discharge from hospital. This will be measured one month after discharge using validated questionnaires (SF 36).
Length of stay at ICU | Participants will be followed for the duration of ICU stay, an expected average of 5 weeks may vary from a few days to several weeks
  To compare whether there is a difference in the length of ICU stay in the standard treatment group versus the intervention group.
time to adminstration of antibiotics (door to needle time) | door to needle time at the ED: from entry at the ED till time to administration of antibiotics
  To compare whether there is a diference in time to administration of antibiotics in the usual care group opposed to baseline measurements prior to start of the trial of the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Prabath WB Nanayakkara, MD, PhD, Principal Investigator — VU Medical Center (VUmc), Amsterdam; P. Stassen, MD, Phd, Principal Investigator — Maastricht Medical Center, Maastricht; E. Oskam, MD, Principal Investigator — Albert Schweitzer Hospital, Dordrecht; H. Nguyen, MD, PhD, Principal Investigator — Maasstad Hospital, Rotterdam
Locations (34):
- Netherlands (34):
  - Amstelland Ziekenhuis, Amstelveen, North Holland
  - Meander Medical Center, Amersfoort
  - Academic Medical Centre, Amsterdam
  - BovenIJ hospital, Amsterdam
  - Onze Lieve Vrouwe Gasthuis Oost (former: St. Lucas Andreas Hospital), Amsterdam
  - Onze Lieve Vrouwe Gasthuis Oost, Amsterdam
  - VU medical center, Amsterdam
  - Rijnstate Hospital, Arnhem
  - Rode Kruis Hospital, Beverwijk
  - Amphia Hospital, Breda
  - Albert Schweitzer Hospital, Dordrecht
  - Gelderse Vallei, Ede
  - Catharina Hospital, Eindhoven
  - Maxima Medical Center, Eindhoven
  - St.Anna Hospital, Geldrop
  - Zuyderland Hospital, Geleen
  - Beatrix Hospital, Gorinchem
  - Spaarne Gasthuis, Haarlem, Haarlem
  - Zuyderland Hospital, Heerlen
  - Elkerliek Hospital, Helmond
  - Spaarne Gasthuis, Hoofddorp
  - Maastricht Medical Center, Maastricht
  - St.Antonius Hospital, Nieuwegein
  - Canisius Wilhemina Hospital, Nijmegen
  - Bravis Hospital, Roosendaal
  - Haven Hospital, Rotterdam
  - Ikazia Hospital, Rotterdam
  - Maasstad Hospital, Rotterdam
  - St.Franciscus Gasthuis, Rotterdam
  - Vlietland Hospital, Schiedam
  - Rivierenland Hospital, Tiel
  - Diakonesse Hospital, Utrecht
  - University Medical Center, Utrecht, Utrecht
  - VieCuri Medical Center, Venlo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ling L, Joynt GM, Lipman J. A narrative review on antimicrobial therapy in septic shock: updates and controversies. Curr Opin Anaesthesiol. 2021 Apr 1;34(2):92-98. doi: 10.1097/ACO.0000000000000954. PMID 33470662
- [Derived] Nannan Panday RS, Lammers EMJ, Alam N, Nanayakkara PWB. An overview of positive cultures and clinical outcomes in septic patients: a sub-analysis of the Prehospital Antibiotics Against Sepsis (PHANTASi) trial. Crit Care. 2019 May 21;23(1):182. doi: 10.1186/s13054-019-2431-8. PMID 31113475
- [Derived] Alam N, Oskam E, Stassen PM, Exter PV, van de Ven PM, Haak HR, Holleman F, Zanten AV, Leeuwen-Nguyen HV, Bon V, Duineveld BAM, Nannan Panday RS, Kramer MHH, Nanayakkara PWB; PHANTASi Trial Investigators and the ORCA (Onderzoeks Consortium Acute Geneeskunde) Research Consortium the Netherlands. Prehospital antibiotics in the ambulance for sepsis: a multicentre, open label, randomised trial. Lancet Respir Med. 2018 Jan;6(1):40-50. doi: 10.1016/S2213-2600(17)30469-1. Epub 2017 Nov 28. PMID 29196046